CLINICAL TRIAL: NCT03772249
Title: A Three-Part, Phase 1, Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics Study of DCR-HBVS in Healthy Volunteers and Patients With Chronic Hepatitis B
Brief Title: Study of Safety and Tolerability of DCR HBVS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dicerna Pharmaceuticals, Inc., a Novo Nordisk company (Industry)
Responsible Party: Sponsor
Organization: Novo Nordisk A/S (Industry)
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: DCR-HBVS-101; U1111-1220-7021 (Other: World Health Organization (WHO))
Record Dates: First submitted 2018-12-03; First posted 2018-12-11 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hepatitis B, Chronic
Keywords: Chronic Hepatitis B; DNA Virus Infections; CHB; HBsAg; Liver Disease; RNAi
MeSH Terms: conditions — Hepatitis B, Chronic; DNA Virus Infections; Liver Diseases

STUDY DESIGN:
Intervention Model Description: Progression from the SAD phase to the first cohort in the MAD phase is contingent upon the Safety Review Committee (SRC) review of a minimum of 14 days post-dose safety and tolerability data from all NHV in at least the first 2 SAD cohorts. The SRC will select one (or more) well-tolerated dose(s) from the SAD phase for administration in the SD and MAD phases. Group B at 3 mg/kg will start in parallel with Group C at the 3 mg/kg dose level. In all study phases, dosing will be staggered with the use of sentinel participants to allow time for the assessment of safety before additional subjects are exposed to study drug. The fixed dosing regimen for Cohorts 4c and 5c was determined following SRC review and assessment of all data up to Cohort 3c. No sentinel dosing will occur in Cohorts 4c and 5c.
Who Masked: Participant, Care Provider, Investigator
Masking Description: This is a double-blind study in which the study site team, the Sponsor, and the participants will be blinded to treatment assignment. The unblinded pharmacist will cover each syringe, prior to transport to the bedside, to ensure blinding. The drug will be injected by an unblinded nurse or physician who is not part of the study team. Participants will be centrally assigned to randomized study intervention using an Interactive Voice/Web Response System (IVRS/IWRS). Cohorts 4c and 5c will be open label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (22):
- Cohort A1 DCR-HBVS (Experimental): Single dose, Subcutaneous injection of 0.1mg/kg of DCR-HBVS (HV)
  Interventions: Drug: DCR-HBVS
- Cohort A1 Placebo (Placebo Comparator): Single dose, Subcutaneous injection of 0.1mg/kg of Placebo for DCR-HBVS (HV)
  Interventions: Drug: Placebo for DCR-HBVS
- Cohort A2 DCR-HBVS (Experimental): Single dose, Subcutaneous injection of 1.5mg/kg of DCR-HBVS (HV)
  Interventions: Drug: DCR-HBVS
- Cohort A2 Placebo (Placebo Comparator): Single dose, Subcutaneous injection of 1.5mg/kg of Placebo for DCR-HBVS (HV)
  Interventions: Drug: Placebo for DCR-HBVS
- Cohort A3 DCR-HBVS (Experimental): Single dose, Subcutaneous injection of 3mg/kg of DCR-HBVS (HV)
  Interventions: Drug: DCR-HBVS
- Cohort A3 Placebo (Placebo Comparator): Single dose, Subcutaneous injection of 3mg/kg of Placebo for DCR-HBVS (HV)
  Interventions: Drug: Placebo for DCR-HBVS
- Cohort A4 DCR-HBVS (Experimental): Single dose, Subcutaneous injection of 6mg/kg of DCR-HBVS (HV)
  Interventions: Drug: DCR-HBVS
- Cohort A4 Placebo (Placebo Comparator): Single dose, Subcutaneous injection of 6mg/kg of Placebo for DCR-HBVS (HV)
  Interventions: Drug: Placebo for DCR-HBVS
- Cohort A5 DCR-HBVS (Experimental): Single dose, Subcutaneous injection of 12mg/kg of DCR-HBVS (HV)
  Interventions: Drug: DCR-HBVS
- Cohort A5 Placebo (Placebo Comparator): Single dose, Subcutaneous injection of 12mg/kg of Placebo for DCR-HBVS (HV)
  Interventions: Drug: Placebo for DCR-HBVS
- Cohort B DCR-HBVS (Experimental): Single dose, Subcutaneous injection of 3mg/kg of for DCR-HBVS (NUC naïve, CHB)
  Interventions: Drug: DCR-HBVS
- Cohort B Placebo (Placebo Comparator): Single dose, Subcutaneous injection of 3mg/kg of Placebo for DCR-HBVS (NUC naïve, CHB)
  Interventions: Drug: Placebo for DCR-HBVS
- Cohort C1 DCR-HBVS (Experimental): 4 doses- Subcutaneous injection of 1.5mg/kg of DCR-HBVS administered every 28 days (NUC experienced, CHB)
  Interventions: Drug: DCR-HBVS
- Cohort C1 Placebo (Placebo Comparator): 4 doses- Subcutaneous injection of 1.5mg/kg of Placebo for DCR-HBVS administered every 28 days (NUC experienced, CHB)
  Interventions: Drug: Placebo for DCR-HBVS
- Cohort C2 DCR-HBVS (Experimental): 4 doses- Subcutaneous injection of 3mg/kg of DCR-HBVS administered every 28 days (NUC experienced, CHB)
  Interventions: Drug: DCR-HBVS
- Cohort C2 Placebo (Placebo Comparator): 4 doses- Subcutaneous injection of 3mg/kg of Placebo for DCR-HBVS administered every 28 days (NUC experienced, CHB)
  Interventions: Drug: Placebo for DCR-HBVS
- Cohort C3 DCR-HBVS (Experimental): 4 doses- Subcutaneous injection of 6mg/kg of DCR-HBVS administered every 28 days (NUC experienced, CHB)
  Interventions: Drug: DCR-HBVS
- Cohort C3 Placebo (Placebo Comparator): 4 doses- Subcutaneous injection of 6mg/kg of Placebo for DCR-HBVS administered every 28 days (NUC experienced, CHB)
  Interventions: Drug: Placebo for DCR-HBVS
- Cohort 4C DCR-HBVS (Experimental): 1 dose- Subcutaneous injection of 100mg (NUC experienced, CHB)
  1 dose- Subcutaneous injection of 200mg (NUC experienced, CHB)
  1 dose- Subcutaneous injection of 400mg (NUC experienced, CHB)
  Interventions: Drug: DCR-HBVS
- Cohort 5C1 DCR-HBVS (Experimental): 4 doses- Subcutaneous injection of 200mg administered every 4 weeks (NUC experienced, CHB)
  Interventions: Drug: DCR-HBVS
- Cohort 5C2 DCR-HBVS (Experimental): 2 doses- Subcutaneous injection of 200mg administered every 8 weeks (NUC experienced, CHB)
  Interventions: Drug: DCR-HBVS
- Cohort 5C3 DCR-HBVS (Experimental): 2 doses- Subcutaneous injection of 400mg administered every 12 weeks (NUC experienced, CHB)
  Interventions: Drug: DCR-HBVS

INTERVENTIONS:
Drug: DCR-HBVS — DCR-HBVS is a synthetic ribonucleic acid interference (RNAi) drug that consists of a double-stranded oligonucleotide conjugated to N-acetyl-D-galactosamine (GalNAc) ligands. DCR-HBVS is a sterile solution of the siRNA (DCR-S219) at a concentration of 195 mg/mL in water for injection (WFI).
  Other Names: DCR-S219
  Arms: Cohort 4C DCR-HBVS; Cohort 5C1 DCR-HBVS; Cohort 5C2 DCR-HBVS; Cohort 5C3 DCR-HBVS; Cohort A1 DCR-HBVS; Cohort A2 DCR-HBVS; Cohort A3 DCR-HBVS; Cohort A4 DCR-HBVS; Cohort A5 DCR-HBVS; Cohort B DCR-HBVS; Cohort C1 DCR-HBVS; Cohort C2 DCR-HBVS; Cohort C3 DCR-HBVS
Drug: Placebo for DCR-HBVS — Sterile 9% saline for injection.
  Other Names: Placebo
  Arms: Cohort A1 Placebo; Cohort A2 Placebo; Cohort A3 Placebo; Cohort A4 Placebo; Cohort A5 Placebo; Cohort B Placebo; Cohort C1 Placebo; Cohort C2 Placebo; Cohort C3 Placebo

SUMMARY:
DCR-HBVS will be evaluated for safety and efficacy in healthy volunteers and chronic hepatitis B patients.

DETAILED DESCRIPTION:
DCR HBVS is being developed for the treatment of chronic hepatitis B (CHB) in adults. The study will be conducted in 3 parts, a single ascending-dose (SAD) phase in normal healthy volunteers (Group A), a single-dose (SD) phase in patients with CHB (Group B), and a multiple ascending-dose (MAD) phase in patients with CHB (Group 1c-3c). Cohort 4c is a single ascending dose with a possible duration of up to 48 weeks. Cohort 5c is a multiple dose cohort with a possible duration of up to 72 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy at the time of screening as determined by medical evaluation.
* Capable of giving informed consent.
* 12-lead ECG within normal limits or with no clinically significant abnormalities.
* Negative screen for alcohol or drugs of abuse.
* Non-smokers for at least 3 months with a negative urinary cotinine concentration at screening.
* BMI within range 18.0 - 32.0 kg/m2 (inclusive).
* Female participants not pregnant, not breastfeeding, and not of childbearing potential or willing to follow contraceptive guidance.
* Chronic hepatitis B infection (Group B and C only).
* Clinical history compatible with compensated liver disease with no evidence of cirrhosis (Group B and C only).
* Continuously on nucleotides (NUC) therapy for at least 12 weeks prior to screening (Group C only).

Exclusion Criteria:

* History of any medical condition that may interfere with the absorption, distribution, or elimination of study drug.
* Poorly controlled or unstable hypertension.
* History of diabetes mellitus treated with insulin or hypoglycemic agents.
* History of asthma requiring hospital admission within the preceding 12 months.
* Evidence of G-6-PD deficiency.
* Currently poorly controlled endocrine conditions, excluding thyroid conditions.
* History of multiple drug allergies or history of allergic reaction to an oligonucleotide or GalNAc.
* Clinically relevant surgical history.
* Use of prescription medications (excluding contraception for women) within 4 weeks prior to the administration of study intervention.
* Use of clinically relevant over-the-counter medication or supplements (excluding routine vitamins) within 7 days of first dosing.
* Has received an investigational agent within the 3 months prior to dosing or is in follow-up of another study.
* Antiviral therapy (other than entecavir or tenofovir) within 3 months of screening or treatment with interferon in the last 3 years (Group B and C only).
* Use within the last 6 months of anticoagulants or systemically administered corticosteroids, immunomodulators, or immunosuppressants (Group B and C only).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2018-12-28 (Actual); Primary Completion 2022-07-12 (Actual); Study Completion 2022-07-12 (Actual)

PRIMARY OUTCOMES:
Number of healthy volunteers with Adverse Events as assessed by CTCAE v5.0 | 4 weeks
  Number of participants with abnormalities in vital signs, electrocardiogram (ECG), and clinically significant laboratory findings
Number participants with non-cirrhotic chronic Hepatitis B with Adverse Events as assessed by CTCAE v5.0 | 16 weeks
  Number of participants with abnormalities in vital signs, electrocardiogram (ECG), and clinically significant laboratory findings

SECONDARY OUTCOMES:
To characterize the pharmacokinetics of DCR-HBVS in healthy volunteers by monitoring plasma pharmacokinetics profiles of DCR-S219 | 4 weeks
  Measure the amount of DCR-HBVS excreted in urine
To characterize the pharmacokinetics of DCR-HBVS in healthy volunteers by monitoring through concentrations of DCR-S219 | 4 weeks
  Measure the amount of DCR-HBVS renal clearance (CLR).
To characterize the pharmacokinetics of DCR-HBVS in participants with non-cirrhotic CHB by monitoring plasma pharmacokinetics profiles of DCR-HBVS. | 12 weeks
  Measure the amount of DCR-HBVS excreted in urine
To characterize the pharmacokinetics of DCR-HBVS in participants with non-cirrhotic CHB by monitoring through concentrations of DCR-HBVS. | 12 weeks
  Measure DCR-HBVS renal clearance (CLR).

OTHER OUTCOMES:
To evaluate the preliminary antiviral efficacy of DCR-HBVS in participants with CHB by monitoring changes in serum HBsAg levels (all Group B and C participants)during and after single dose and 12 weeks of treatment with DCR HBVS. | 12 weeks
  Proportion of participants achieving at least a 1-log reduction in HBsAg AND achieving a HBsAg level < 100 IU/mL at last scheduled visit Time to HBsAg loss (Kaplan-Mayer) Time to anti-HBs seroconversion
To evaluate the preliminary antiviral efficacy of DCR-HBVS in participants with CHB by monitoring HBeAg levels (HBeAg+ participants only) during and after single dose and 12 weeks of treatment with DCR HBVS. | 12 weeks
  % of participants with HBeAg loss and anti HBe at last scheduled visit (if HBeAg positive at study entry)
To evaluate the preliminary antiviral efficacy of DCR-HBVS in participants with CHB by monitoring HBV DNA levels (all Group B and C participants) during and after single dose and 12 weeks of treatment with DCR HBVS. | 12 weeks
  Proportion of participants achieving HBV DNA < 2000 IU/mL (if > 2,000 IU/mL at Baseline); and proportion of participants achieving PCR-nondetectable HBV DNA (if HBV DNA was detectable at Baseline).
To characterize the pharmacodynamics (PD) of DCR-HBVS on plasma levels of HBsAg and HBV in blood. | 12 weeks
  Track post-treatment duration of any observed efficacy effects.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Bowman, MD, Study Director — Dicerna Pharmaceuticals
Locations (9):
- Australia (2):
  - Monash Health, Clayton, Victoria
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
- Queen Mary Hospital (The University of Hong Kong), Hong Kong, Hong Kong
- New Zealand (2):
  - Clinical Site, Auckland
  - Middlemore Hospital, Auckland
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Seoul Metropolitan Government - Seoul National University Boramae Medical Center, Soeul
- Thailand (2):
  - King Culalongkorn Memorial Hospital, Bangkok
  - Srinagarind Hospital, Khon Kaen

REFERENCES:
- [Derived] Gane EJ, Kim W, Lim TH, Tangkijvanich P, Yoon JH, Sievert W, Sukeepaisarnjaroen W, Thompson AJ, Pavlovic V, Surujbally B, Wat C, Brown BD, Achneck HE, Yuen MF. First-in-human randomized study of RNAi therapeutic RG6346 for chronic hepatitis B virus infection. J Hepatol. 2023 Nov;79(5):1139-1149. doi: 10.1016/j.jhep.2023.07.026. Epub 2023 Jul 29. PMID 37524230